CLINICAL TRIAL: NCT05690893
Title: Evaluation of the Physiological Crystalline Lens Tilt Using Longitudinal and High-resolution Swept-source Optical Coherence Tomography: a Retrospective Study
Brief Title: Crystalline Lens Tilt Evaluation Using Swept-source Optical Coherence Tomography
Acronym: PhysTilt
Status: Completed | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Other Study IDs: KUK-Ophthalmology-010
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Cataract Surgery
Keywords: Cataract; CASIA2; IOL Master700
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this retrospective study is to quantify the physiological lens tilt of the phakic eye.

The main question it aims to answer is:

-What influence does misalignment or tilting of IOLs have on visual quality?

Preoperative biometry data are compared with anterior segement OCT data.

Measurements were obtained using high-resolution swept-source optical coherence tomography. The influence of biometric measurements on tilt is analyzed.

DETAILED DESCRIPTION:
The human (crystalline or phakic) lens is located in the capsular bag which is attached to zonules. Zonules are fibres, that hold the lens in place. In the course of life, an opacification on the lens occurs, which is called cataract. To replace the cloudy lens, cataract surgery is being performed and an artificial intraocular lens (IOL) is implanted in the eye, after the phakic lens is removed. Misalignment or tilting of IOLs can result in reduction of visual quality, therefore prediction of the position may be beneficial. Modern optical coherence tomography (OCT) devices already provide profound information about phakic lens tilt. Still there is little data on the values that influence the tilt of the crystalline lens. Before each cataract surgery, each eye is measured using biometry (IOL Master 700). However, a statement about the tilt cannot be made on the basis of the results of IOL Master 700. For this purpose, an anterior segment OCT is required (CASIA 2). In this study, preoperative biometry data are compared with anterior segment OCT data. A statistical analysis will then be performed to identify the biometric parameters that can predict phakic lens tilt.

ELIGIBILITY:
Inclusion Criteria:

* Planned cataract surgery in one or both eyes
* Minimum age of 21 years

Exclusion Criteria:

* Opacities of the refracting media
* Measurement error in the context of preliminary investigation
* pseudophakia

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 21 and 100 years who received preliminary examinations as part of cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Physiological lens tilt | June 2020 - October 2022
  SS-OCT measurements (IOLMaster700 and Casia2) to investigate axial eye length, anterior chamber depth and lens thickness and their influence on lens tilt

SECONDARY OUTCOMES:
Correlation of biometric data | June 2020 - October 2022
  Correlation of other biometric data (lens thickness, anterior chamber depth, white-to-white) with lens tilt

CONTACTS AND LOCATIONS:
Overall Officials: Nino Hirnschall, MD, Principal Investigator — Johannes Kepler University
Locations (1):
- Johannes Kepler University Linz, Linz, Upper Austria, Austria